CLINICAL TRIAL: NCT00001477
Title: Monitoring Patients for Developing Communicable and Opportunistic Infections and for Responding to Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950176; 95-I-0176
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Communicable Diseases; Opportunistic Infections
Keywords: Communicable Infection; Monitoring; Non-Invasive Tests; Opportunistic Infection
MeSH Terms: conditions — Communicable Diseases; Opportunistic Infections

SUMMARY:
Patients are exposed to infectious agents regularly, regardless of their immunologic status. Traditionally clinicians have decided to institute prophylaxis based on epidemiologic factors, skin test (i.e. PPD), or immunologic parameters. A quantitative and specific method that is non-invasive, such as quantitative PCR, would be desirable to more precisely define those who would benefit from prophylaxis. Similarly, when patients develop disease and are being treated, quantitative, non-invasive techniques are needed to assess response to therapy. This project is designed to develop and test quantitative tests using blood, urine, or sputum samples.

DETAILED DESCRIPTION:
Patients are exposed to infectious agents regularly, regardless of their immunologic status. Traditionally clinicians have decided to institute prophylaxis based on epidemiologic factors, skin test (i.e. PPD), or immunologic parameters. A quantitative and specific method that is non-invasive, such as quantitative PCR, would be desirable to more precisely define those who would benefit from prophylaxis. Similarly, when patients develop disease and are being treated, quantitative, non-invasive techniques are needed to assess response to therapy. This project is designed to develop and test quantitative tests using blood, urine, or sputum samples.

ELIGIBILITY:
Patients older than 18 years of age.

Ability to give informed consent.

No medical contraindication to phlebotomy.

Epidemiologically at risk for tuberculosis or for an opportunistic infection.

Patients who can identify a responsible health care provider as someone willing to provide clinical information and to receive medically important information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1995-08; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Drouet E, Colimon R, Michelson S, Fourcade N, Niveleau A, Ducerf C, Boibieux A, Chevallier M, Denoyel G. Monitoring levels of human cytomegalovirus DNA in blood after liver transplantation. J Clin Microbiol. 1995 Feb;33(2):389-94. doi: 10.1128/jcm.33.2.389-394.1995. PMID 7714198
- [Background] Patel R, Smith TF, Espy M, Wiesner RH, Krom RA, Portela D, Paya CV. Detection of cytomegalovirus DNA in sera of liver transplant recipients. J Clin Microbiol. 1994 Jun;32(6):1431-4. doi: 10.1128/jcm.32.6.1431-1434.1994. PMID 8077384
- [Background] Spector SA, Merrill R, Wolf D, Dankner WM. Detection of human cytomegalovirus in plasma of AIDS patients during acute visceral disease by DNA amplification. J Clin Microbiol. 1992 Sep;30(9):2359-65. doi: 10.1128/jcm.30.9.2359-2365.1992. PMID 1328287